CLINICAL TRIAL: NCT01158456
Title: Mechanisms of Ethnic/Racial Differences in Lung Cancer Due to Cigarette Smoking: Project 5: Metabolism of NNK Among African Americans
Brief Title: Metabolism of NNK Among African Americans
Acronym: Project 5
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010NTLS056; 1P01CA138338-01A1 (NIH)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: smoking; lung cancer; ethnic racial differences; tobacco specific nitrosamines; metabolism of carcinogens
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sample (approximately 40 ml) will be drawn from each study participant at the baseline visit. Approximately 33 ml will be used immediately for the study, and the remaining two 3-ml volumes will be reserved for future use. The various components of the blood including buffy coat (white blood cells), red blood cells, plasma, and serum will be separated immediately after their collection, labelled using a unique subject number, and stored in a -80C freezer. Urine samples and oral cells will be collected from study subjects at various time points. All these samples will be labelled using a unique subject number, and stored at a -80C freezer.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- African Americans: Subjects will be classified as African American if they report themselves, biological parents and both sets of biological grandparents as African American or African descent.
- European American: Subjects will be classified as European American if they report themselves, biological parents and both sets of biological grandparents as European American or European descent.

SUMMARY:
Metabolism and DNA adduct formation are critical in cancer induction by NNK. The investigators goal is to understand whether the observed ethnic/racial differences in lung cancer incidence are due to variations in NNK metabolism. The investigators overall hypothesis is that cancer susceptibility relates to carcinogen dose and to the balance between carcinogen metabolic activation and detoxification. The investigators propose to test this hypothesis via investigation of potential differences in NNK metabolic activation and detoxification in African American and European American smokers.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death in the United States, with the annual number of cases estimated at 162,460 deaths per year. It is more prevalent in African Americans as compared to European Americans. Cigarette smoking causes up to 90% of lung cancer, being the major risk factor in both African Americans and European Americans.

Tobacco-specific nitrosamines (TSNA) are among the most significant carcinogens in tobacco products. Multiple international studies clearly document the occurrence of substantial amounts of these carcinogens in both unburned tobacco and tobacco smoke. One of the most prevalent of these compounds, 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), is present in both unburned tobacco and cigarette smoke, and is a remarkably effective lung carcinogen in laboratory animals, inducing lung tumors in rodents independent of the route of administration. 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), a metabolite of NNK, is also a pulmonary carcinogen. NNK has been classified by the International Agency for Research on Cancer as a Group 1 carcinogen (carcinogenic to humans). Consistent with this, 2 recent studies by our group have demonstrated that levels of NNAL in serum or urine are related to lung cancer in smokers.

Our primary aim is to conduct a comprehensive analysis of urinary biomarkers of NNK metabolic activation and detoxification in African American and European American smokers. We hypothesize that, after adjustment for smoking level, the relative contribution of the biomarkers of NNK metabolic activation to the total amount of NNK metabolites will be higher in African Americans as compared to European Americans. Our secondary aim is to measure in exfoliated oral mucosa cells of African American and European American smokers DNA adducts formed as a result of NNK metabolic activation. The results of these measurements will offer a direct measure of NNK-induced DNA damage in smokers, and will be critical to an understanding of the balance between the urinary excretion of NNK metabolites and the extent of NNK DNA binding. We hypothesize that African Americans will have in the DNA of their oral mucosa cells higher levels of NNK-derived DNA adducts as compared to European Americans. Finally, we will investigate the relationship between levels of NNK-derived DNA adducts measured in oral mucosa cells and the rates of repair of these adducts in cultured lymphocytes from our subjects. These measurements will allow us to evaluate more fully the role of variations in NNK metabolism in the observed differences in lung cancer risk between European American and African American smokers. We expect that that African Americans will have lower capacity to repair NNK-induced DNA damage as compared to European Americans, and this will correlate with higher levels of NNK-derived buccal DNA adducts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with a smoking history of at least 10 cigarettes daily for at least 1 year;
2. Subjects report themselves, biological parents and both sets of biological grandparents as

   * African American or African descent or
   * European American or European descent
3. Subjects are in apparently good physical health (no unstable medical condition)
4. Subjects are in stable, good mental health (e.g. not currently, within the past 6 months, experiencing unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the PRIME-MD);
5. Subjects have provided written informed consent to participate in the study.

Exclusion Criteria:

1. Unstable medical conditions including cancer, coronary heart disease and arrhythmia
2. Cannot or unwilling to identify ethnic/racial ancestry
3. Women who are currently pregnant or breast feeding
4. Currently using any other tobacco or nicotine-containing product
5. Currently taking any medications that affect relevant metabolic enzymes.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be classified as African American if they report themselves, biological parents and both sets of biological grandparents as African American or African descent. Similar criteria will be applied to European Americans (e.g., self, both parents and four grandparents of European American or European descent). Subjects will be evenly divided by gender.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Conduct a comprehensive analysis of urinary biomarkers of NNK metabolic activation and detoxification in African American and European American smokers. | 10 days
  We will recruit smokers to smoke specially prepared cigarettes containing [pyridine-D4]NNK, and measure deuterium-labeled NNK metabolites in the urine of these subjects. The rationale for the use of deuterium-labeled NNK is that we need to specifically identify NNK-derived metabolites, because these biomarkers are also formed as a result of nicotine metabolism. Our overall hypothesis is that the relative contribution of the biomarkers of NNK metabolic activation to the total amount of NNK metabolites will be higher in African Americans as compared to European Americans.

SECONDARY OUTCOMES:
Measure in exfoliated oral mucosa cells of African American and European American smokers DNA adducts formed as a result of NNK metabolic activation. | 10 days
  We will collect exfoliated oral mucosa cell samples from the recruited subjects. DNA isolated from these samples will be analyzed for [pyridine-D4]NNK-derived adducts. Our overall hypothesis in this Specific Aim is that African Americans will have in the DNA of their oral mucosa cells higher levels of NNK-derived DNA adducts as compared to European Americans.
Assess the repair of NNK-induced DNA damage. | 10 days
  We will investigate the relationship between the levels of NNK-derived DNA adducts measured in the oral mucosa cells and the rates of repair of these adducts in cultured lymphocytes from our subjects. Our overall hypothesis for this Specific Aim is that African Americans will have lower capacity to repair NNK-induced DNA damage as compared to European Americans, and this will correlate with higher levels of [pyridine-D4]NNK-derived buccal DNA adducts.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Tobacco Research Programs University of Minnesota, Minneapolis, Minnesota, United States